CLINICAL TRIAL: NCT04734964
Title: Effect of Two Types of Exercise Training on Fine Motor Skills in Adolescents: Association With Testosterone
Brief Title: Effect of Exercise Training on Fine Motor Skills
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lithuanian Sports University (Other)
Collaborators: Medical School Hamburg (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: LithuanianSportsU-5
Record Dates: First submitted 2021-01-25; First posted 2021-02-02 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Fine Motor Skills; Testosterone Concentration
Keywords: school, cardiovascular exercise, coordinative exercise
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (No Intervention): Participants underwent only common physical education classes twice per week for 45 minutes each and no additional after-school exercises.
- Coordinative exercise group (Experimental): Participants had common physical education classes twice per week for 45 minutes each, and additional exercise sessions were held three times per week for 45 minutes after school.
  Interventions: Behavioral: exercise training
- Cardiovascular exercise group (Experimental): Participants had common physical education classes twice per week for 45 minutes each, and additional exercise sessions were held three times per week for 45 minutes after school.
  Interventions: Behavioral: exercise training

INTERVENTIONS:
Behavioral: exercise training — Exercise training session for 45 minutes.
  Arms: Cardiovascular exercise group; Coordinative exercise group

SUMMARY:
Despite the importance of physical activity for adolescent physical development, the specific impact of different types of exercise training on fine motor skills and testosterone concentration is unknown. A primary aim of this study was to analyze the benefits of cardiovascular and coordinative exercise training on fine motor skills in an adolescent population. A second aim of our study was to determine the testosterone concentration after physical stress of cardiovascular and coordinative exercise training and if testosterone was related to fine motor skills among adolescents following an exercise training intervention.

DETAILED DESCRIPTION:
We assigned 135 adolescents (68 girls, 12-15 years of age) from Lithuania. Adolescents were assigned to one of three groups: control group (CON) (n = 46; 23 girls), coordinative exercise (CE) (n = 41; 22 girls), and cardiovascular exercise (CVE) group (n = 48; 23 girls). Participants performed all necessary tests according to the study protocol one week before the intervention. Adolescents were familiarized with the tests on a separate day before the first assessment. A second set of tests was performed one week after the 10-week exercise intervention.

The exercise intervention period was 10 weeks. Exercises were led by a Physical Education teacher. Experimental groups had common physical education classes twice per week for 45 minutes each, and additional exercise sessions were held three times per week for 45 minutes after school.

ELIGIBILITY:
Inclusion Criteria:

* absence of physical impairment (e.g. traumatic injury)
* absence of mental impairment (e.g. mental retardation)
* no consumption of psychotropic medications

Exclusion Criteria:

• restrictions to do exercises (based on Medical certificate issued by the Physician)

Ages: 12 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 135 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-09-28 (Actual)

PRIMARY OUTCOMES:
Fine motor skills assessed by the Flower trail test | baseline and week 10
  Flower trail test was used to assess fine motor skills. The participant has to draw a line between two solid lines as accurately as possible and without lifting a pen. A higher score in the flower trail test means more mistakes made. Change = (week 10 score - baseline score)
Salivary testosterone concentration | baseline and week 10
  Hormone concentration within the saliva sample was measured using the enzyme-linked immunosorbent assay (IBL, Hamburg, Germany). Change = (week 10 score - baseline score).

SECONDARY OUTCOMES:
Hand-eye coordination assessed by the Hand-eye coordination test | baseline and week 10
  Participant has to throw a tennis ball against a wall and catch and repeat this for 30 seconds. A number of successful catches is recorded, higher score shows better coordination. Change = (week 10 score - baseline score).
static balance assessed by the Flamingo balance test | baseline and week 10
  Flamingo balance test is used to assess static balance. Every attempt to maintain balance for 1 minute is counted as a score. Small values (closer to 1) indicate a better balance. Change = (week 10 score - baseline score)
Cardiorespiratory fitness assessed by the Shuttle Run Test | baseline and week 10
  On this test, the participant must run back and forth between two lines (20 meters apart) with increasing intensity. Higher score means a better cardiorespiratory fitness. Change = (week 10 score - baseline score).

CONTACTS AND LOCATIONS:
Overall Officials: Juste Knatauskaite, Principal Investigator — Lithuanian Sports University
Locations (1):
- Lithuanian Sports University, Kaunas, Lithuania

IPD SHARING:
Plan to Share IPD: No